CLINICAL TRIAL: NCT02465333
Title: Fat Grafting and Retention for Heel Fat Pad Atrophy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Jeffrey A. Gusenoff, MD, Associate Professor of Surgery, University of Pittsburgh
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: PRO14110358
Record Dates: First submitted 2015-05-27; First posted 2015-06-08 (Estimated); Last update posted 2024-01-31 (Actual); Status verified 2024-01

CONDITIONS: Heel Fat Pad Atrophy
Keywords: heel; atrophy; fat; adipose tissue; fat pad
MeSH Terms: conditions — Atrophy; Platelet Glycoprotein IV Deficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pathway A (Other): Screening visit followed by heel fat grafting procedure with local anesthetic and visits at:
  1 week Post op study visit 2 (1 month) Post op study visit 3 (2 month) Post op study visit 4 (6 month) Post op study visit 5 (12 month) Crossover to standard podiatry visits Study visit 6 (18 months) Study visit 7 (24 months)
  Interventions: Procedure: Heel Fat Grafting
- Pathway B (Other): Screening visit followed by:
  Study visit 1 (6 months) Study Visit 2 (12 months) Crossover to Pathway A
  Heel fat grafting procedure and local anesthetic and visits at:
  1 week Post op study visit 2 (1 month post procedure) Post op study visit 3 (2 month post procedure) Post op study visit 4 (6 month post procedure) Post op study visit 5 (12 month post procedure)
  Interventions: Procedure: Heel Fat Grafting

INTERVENTIONS:
Procedure: Heel Fat Grafting — Fat grafting is widely used by plastic surgeons and is considered a standard of care procedure in plastic surgery. Fat tissue to be used for grafting is harvested with a small liposuction cannula. The fat is then centrifuged, cleaned, and loaded into 1cc syringes and injected into the heel fat pad using specialized cannulas.
  Postoperatively, the foot will be bandaged for twenty-four hours and the subject will be advised to limit ambulation. Over the next three weeks, the patient will be instructed to wear a cushioned, supportive sneaker and participate in only activities of normal daily living, with no excessive aerobic activity.

SUMMARY:
Plantar heel pain is the most common problem of the foot. Plantar fasciitis is the leading cause of this pain, accounting for 11-15% of all foot symptoms seeking professional care, and occurs in 10% of the US population. The cause of heel pain can be from bone, soft tissue, nerve, or systemic disease. The second most common cause of heel pain is fat pad atrophy, followed by a combination of both fat pad atrophy and plantar fasciitis. [1-4] Fat pad displacement may be seen in the heel as well.

Current treatments for plantar fasciitis include stretching and external support with orthotics with the goal of reducing local pressure as well as tissue breakdown.[5] However, patient compliance with extrinsic devices is challenging, and they may experience increased friction, irritation and breakdown at a different location on the foot due to thickness of the device in the shoe. Also, the patient must replace the device as soon as it breaks down but the breakdown often goes unnoticed. Failure of conservative management may lead to treatment with steroids or surgical intervention by endoscopic plantar fasciotomy, open fasciotomy or excision of bone spurs. Injection of steroids can instigate or exacerbate pre-existing heel fat pad atrophy. Autologous fat grafting to the heel may reduce plantar pressures, and thus serve as a treatment for heel pain. Autologous fat grafting is currently under investigation for a myriad of clinical scenarios.[6-19] Even though autologous fat grafting is not yet an established therapeutic approach for the cited indications, some of the reported results have been intriguing.[19] The variable resorption of fat, however, is an important confounding factor in all these studies. Currently the literature reports fat retention rates ranging from 25% to 80%.[20]

The specific aim of this study is to assess the adipose stem cell characteristics in patients undergoing autologous fat grafting for heel fat pad atrophy and correlate these characteristics with fat retention. Data from this study will help determine the characteristics of the adipose stem cells in this population and open the door to additional studies. This pilot study will also help build new collaborative efforts between Foot and Ankle Specialists, Plastic Surgery, and Adipose Stem Cell Biologists, combining biomechanical expertise with fat grafting and basic science expertise.

DETAILED DESCRIPTION:
With the growth of the investigators diabetic and geriatric populations today, greater demand is being placed on the medical arena to treat their complications. There is currently no effective treatment for diabetic neuropathy which is one of the leading reasons for the development of diabetic ulcerations with high peak plantar pressure. An optical pedobarograph has been used to help study the pressures under the foot.[24] By minimizing high peak plantar pressures through autologous fat transfer, pain and skin lesions have the potential to be minimized.

Restoring the plantar fat pad with autologous fat grafting has the potential to improve foot function, decrease foot pain, bone pain, and nerve pain in the sensate foot and potentially decrease the incidence of foot ulceration in diabetics. It also serves to increase shock absorption during gait. Research has shown greater viability and cellular function with fat grafts processed using the Coleman technique than with other techniques.[25] It is the investigators aim to implement the Coleman technique to increase pedal shock absorption on a long term basis. Increasing shock absorption is prophylactic for reducing calcaneal contusions and stress fractures. By limiting an antalgic, compensatory gait, this will limit injury to the patient's superstructure and/or the contralateral foot and leg, ultimately improving the patient's overall systemic health.

By minimizing high peak plantar pressures through autologous fat transfer, more severe diabetic complications may be minimized. Heel fat pad augmentation may reduce ulcer formation and/or reformation, and reduce the subsequent comorbid conditions of osteomyelitis and amputation. Typically, ulceration due to bone prominence may be best treated by surgical resection of the prominent bone. However, there exists a population of diabetics that will have a greater chance of developing an acute Charcot event post-surgery or transfer lesions that will ultimately break down. Transfer lesions and re-ulceration is considered a common complication after diabetic foot ulcer surgery.[26] Also some patients may not be medically stable making an aggressive osseous surgical procedure inadvisable. If autologous fat grafting does prove to be effective in the foot, it could become a concomitant procedure performed with osseous procedures for a target population of diabetics to limit transfer lesions and ulceration post operatively.

If the proposed aims are achieved, patients will be able to have long lasting reconstruction of the heel fat pad with a minimally invasive procedure using autologous tissue. The ultimate costs of maintaining specialized extrinsic padding, shoe gear, and issues with patient compliance can be reduced or eliminated. It could potentially save the medical arena the costs of treating diabetic ulcerations and the resultant complications. The need for other fillers such as silicone which can migrate and involve lymph nodes can be eliminated, as can the need for repeat injections of other temporary fillers which are currently used without any evidence-based medicine. This project will improve scientific knowledge, technical capability, and clinical practice in both the field of plastic surgery and podiatry. Not only will it influence these fields, but augmenting the heel fat pad has the potential to benefit diabetics, geriatric patients, Wounded Warriors with amputations whom have differential loading of their remaining lower extremity, athletes, and cosmetic patients who would like a more active lifestyle than their current foot pain allows.

Determining the intrinsic fat properties that lead to a consistent and high fat retention rate can have an enormous impact on the current clinical field of fat grafting. Over 80,000 autologous fat grafting procedures were documented in 2013 by The American Society for Aesthetic Plastic Surgery.[27] Determining the factors related to fat retention can aid surgeons in determining the potential amount of fat that may be necessary for optimizing retention, and potentially avoid need for recurrent treatments. Further on, this data would also allow bioengineers to specifically develop fillers using the constituents known to be of importance for the final retention. This project will increase scientific knowledge, technical capability, and improve clinical collaboration between Foot and Ankle Specialists, Plastic Surgeons, and Adipose Stem Cell Biologists.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or older and able to provide informed consent
* Patients with foot pain at the plantar surface of the foot near the head of the metacarpals
* 6 months post any surgical intervention to the foot
* Willing and able to comply with follow up examinations, including ultrasounds and pedobarographic studies

Exclusion Criteria:

* Age less than 18 years
* Inability to provide informed consent
* Feet with open ulcerations or osteomyelitis
* Poorly controlled Diabetics with hemoglobinA1C > 7.
* Active infection anywhere in the body
* Diagnosed with cancer within the last 12 months and /or presently receiving chemotherapy or radiation treatment
* Known coagulopathy
* Systemic disease that would render the fat harvest and injection procedure, along with associated anesthesia, unsafe to the patient.
* Pregnancy
* Subjects with a diagnosis of Schizophrenia or Bipolar Disorder (Subjects who are found to be stable on medication and receive psychiatric clearance could be eligible for study participation per the Physician's discretion).
* Tobacco use: Last use within 1 year per patient report

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2015-05; Primary Completion 2021-06 (Actual); Study Completion 2021-07 (Actual)

PRIMARY OUTCOMES:
Pedobarograph to measure foot pressure | baseline and 2 years
  Change in foot pressure will be measured on the pedobarograph in kg/cm2 or psi. These measures will be performed before and after treatment with fat grafting to assess changes over time.

SECONDARY OUTCOMES:
Adipose stem cell counts | baseline and 2 years
  Extra fat from the liposuction procedure will be sent for adipose stem cell analysis to correlate to retention of the fat over time.
Ultrasound to measure tissue thickness | baseline 2 years
  Tissue thickness will be measured by ultrasound as mm. These measures will be performed before and after treatment with fat grafting to assess changes over time.
Manchester Foot Disability Index for pain | baseline and 2 years
  Pain will be evaluated with the Manchester Foot Disability Index.These measures will be performed before and after treatment with fat grafting to assess changes over time.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey A Gusenoff, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- UPMC Department of Plastic Surgery, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bowling FL, Metcalfe SA, Wu S, Boulton AJ, Armstrong DG. Liquid silicone to mitigate plantar pedal pressure: a literature review. J Diabetes Sci Technol. 2010 Jul 1;4(4):846-52. doi: 10.1177/193229681000400412. PMID 20663447
- [Background] Abouaesha F, van Schie CH, Armstrong DG, Boulton AJ. Plantar soft-tissue thickness predicts high peak plantar pressure in the diabetic foot. J Am Podiatr Med Assoc. 2004 Jan-Feb;94(1):39-42. doi: 10.7547/87507315-94-1-39. PMID 14729989
- [Background] Abouaesha F, van Schie CH, Griffths GD, Young RJ, Boulton AJ. Plantar tissue thickness is related to peak plantar pressure in the high-risk diabetic foot. Diabetes Care. 2001 Jul;24(7):1270-4. doi: 10.2337/diacare.24.7.1270. PMID 11423514
- [Background] Boulton AJ, Franks CI, Betts RP, Duckworth T, Ward JD. Reduction of abnormal foot pressures in diabetic neuropathy using a new polymer insole material. Diabetes Care. 1984 Jan-Feb;7(1):42-6. doi: 10.2337/diacare.7.1.42. PMID 6546713
- [Background] Young MJ, Cavanagh PR, Thomas G, Johnson MM, Murray H, Boulton AJ. The effect of callus removal on dynamic plantar foot pressures in diabetic patients. Diabet Med. 1992 Jan-Feb;9(1):55-7. doi: 10.1111/j.1464-5491.1992.tb01714.x. PMID 1551311
- [Background] Chairman EL. Restoration of the plantar fat pad with autolipotransplantation. J Foot Ankle Surg. 1994 Jul-Aug;33(4):373-9. PMID 7951190
- [Background] van Schie CH, Whalley A, Armstrong DG, Vileikyte L, Boulton AJ. The effect of silicone injections in the diabetic foot on peak plantar pressure and plantar tissue thickness: a 2-year follow-up. Arch Phys Med Rehabil. 2002 Jul;83(7):919-23. doi: 10.1053/apmr.2002.33058. PMID 12098150
- [Background] Pu LLQ, Coleman SR, Cui X, Ferguson REH Jr, Vasconez HC. Autologous fat grafts harvested and refined by the Coleman technique: a comparative study. Plast Reconstr Surg. 2008 Sep;122(3):932-937. doi: 10.1097/PRS.0b013e3181811ff0. PMID 18766062
- [Background] Kwan RL, Zheng YP, Cheing GL. The effect of aging on the biomechanical properties of plantar soft tissues. Clin Biomech (Bristol). 2010 Jul;25(6):601-5. doi: 10.1016/j.clinbiomech.2010.04.003. Epub 2010 May 8. PMID 20457479
- [Background] Veves A, Boulton AJ. The optical pedobarograph. Clin Podiatr Med Surg. 1993 Jul;10(3):463-70. PMID 8364849
- [Background] Walter Stephen Snyder 1909-1977. Health Phys. 1978 Jan;34(1):1-2. No abstract available. PMID 340428
- [Background] Balkin SW. Injectable silicone and the foot: a 41-year clinical and histologic history. Dermatol Surg. 2005 Nov;31(11 Pt 2):1555-9; discussion 1560. doi: 10.2310/6350.2005.31241. PMID 16416638
- [Background] van Schie CH, Whalley A, Vileikyte L, Wignall T, Hollis S, Boulton AJ. Efficacy of injected liquid silicone in the diabetic foot to reduce risk factors for ulceration: a randomized double-blind placebo-controlled trial. Diabetes Care. 2000 May;23(5):634-8. doi: 10.2337/diacare.23.5.634. PMID 10834422
- [Background] Nicoletti G, Brenta F, Jaber O, Laberinti E, Faga A. Lipofilling for functional reconstruction of the sole of the foot. Foot (Edinb). 2014 Mar;24(1):21-7. doi: 10.1016/j.foot.2014.02.003. Epub 2014 Mar 6. PMID 24656457
- [Background] Hsu CC, Tsai WC, Hsiao TY, Tseng FY, Shau YW, Wang CL, Lin SC. Diabetic effects on microchambers and macrochambers tissue properties in human heel pads. Clin Biomech (Bristol). 2009 Oct;24(8):682-6. doi: 10.1016/j.clinbiomech.2009.06.005. Epub 2009 Jul 19. PMID 19619918
- [Background] Hsu CC, Chen CP, Lin SC, Tsai WC, Liu HT, Lin YC, Lee HJ, Chen WP. Determination of the augmentation effects of hyaluronic acid on different heel structures in amputated lower limbs of diabetic patients using ultrasound elastography. Ultrasound Med Biol. 2012 Jun;38(6):943-52. doi: 10.1016/j.ultrasmedbio.2012.02.031. Epub 2012 Apr 12. PMID 22502884
- [Background] Stupar M, Tibbles A. Heel pain and HIV-associated lipodystrophy: a report of two cases. J Can Chiropr Assoc. 2008 Jun;52(2):103-9. PMID 18516231
- [Background] Campanelli V, Fantini M, Faccioli N, Cangemi A, Pozzo A, Sbarbati A. Three-dimensional morphology of heel fat pad: an in vivo computed tomography study. J Anat. 2011 Nov;219(5):622-31. doi: 10.1111/j.1469-7580.2011.01420.x. Epub 2011 Aug 17. PMID 21848602
- [Background] Yi TI, Lee GE, Seo IS, Huh WS, Yoon TH, Kim BR. Clinical characteristics of the causes of plantar heel pain. Ann Rehabil Med. 2011 Aug;35(4):507-13. doi: 10.5535/arm.2011.35.4.507. Epub 2011 Aug 31. PMID 22506166
- [Background] Uzel M, Cetinus E, Ekerbicer HC, Karaoguz A. Heel pad thickness and athletic activity in healthy young adults: a sonographic study. J Clin Ultrasound. 2006 Jun;34(5):231-6. doi: 10.1002/jcu.20230. PMID 16673365